CLINICAL TRIAL: NCT00501865
Title: An Open, Randomised, Two-period Crossover Study to Investigate the Effect of Food on the Pharmacokinetics of GW273225 Administered Immediately After Food and Administered in Fasted State to Healthy Male and Female Subjects
Brief Title: Study to Assess the Effect of Food on the Concentration of GW273225 in the Body of Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NAP109169
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Bipolar Disorder
Keywords: healthy volunteers; food effect,; quantitative pharmacokinetic analysis,; GW273225,
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): Subjects will be randomized to sequence AB, where A represents fasted state and B represents fed state. Subjects will be administered a single oral dose of GW273225 50 milligrams (mg) in the fasted state in dosing period 1. The subjects will receive a single oral dose of GW273225 50 mg immediately after a high fat breakfast in dosing period 2. There will be at least 21 days between doses for the fasted and fed treatment phases of the study.
  Interventions: Drug: GW273225
- Sequence BA (Experimental): Subjects will be randomized to sequence BA, where A represents fasted state and B represents fed state. Subjects will be orally administered a single dose of GW273225 50 mg immediately after a high fat breakfast in dosing period 1. The subjects will receive a single oral dose of GW273225 50 mg in the fasted state in dosing period 2. There will be at least 21 days between doses for the fed and fasted treatment phases of the study.
  Interventions: Drug: GW273225

INTERVENTIONS:
Drug: GW273225 — GW273225 will be available as white tablets containing 25 mg GW273225.The study drug will be taken with 240 milliliters of water at room temperature.

SUMMARY:
The rationale of this study is to assess whether or not food affects the absorption of GW273225 into the blood of healthy male and female volunteers in order to evaluate whether or not this drug should be given at a certain time relative to the consumption of food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged 18-55 years, inclusive.
* Body weight 45-100kg and BMI 19-29.9 kg/m2 inclusive.
* Post-menopausal females (longer than two years). Or Pre-menopausal females with a documented hysterectomy and/or bilateral oophorectomy, the latter only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Female subjects of child bearing potential willing to participate commit to use a double-barrier method of contraception. One of the following methods is acceptable as the sole method of contraception if there is indisputable data that it is >99% effective, otherwise it should be used with a barrier method (condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicidal foam/gel/film/cream/suppository): Documented tubal ligation. Documented placement of an IUD or IUS. Male partner sterilisation prior to the female subject's entry into the study and is the sole partner for that female subject.
* No abnormality on relevant clinical examination or clinical chemistry or haematology examination at the pre-study medical examination.
* A normal 12-lead ECG at the pre-study medical examination
* A negative pre-study Hepatitis B, Hepatitis C, and HIV antibody result at screening.
* A negative pre-study urine drug screen.
* A negative screen for alcohol.
* Subjects must smoke <10 cigarettes per day.
* The subject is able to understand and comply with the study and it's restrictions.

Exclusion Criteria:

* An unwillingness of the male subject to use a double-barrier method of contraception.
* Female subject is pregnant or lactating.
* Female subjects using hormonal contraceptive precautions including progesterone-coated IUD and oral contraceptives.
* Female subjects using hormonal replacement therapy.
* History of alcohol/drug abuse or dependence within 12 months of the study
* The subject has a positive pre-study urine drug/ urine alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Weekly alcohol intake of more than 21 units or an average daily intake of greater than three units (for male subjects) or weekly alcohol intake more than 14 units or an average daily intake of greater than two units (for female subjects).
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* History of sensitivity to any of the study medications, or components thereof.
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.
* History of hypersensitivity to lamotrigine or GW273225.
* History of clinically relevant skin rashes and allergies that, in the opinion of the investigator, might interfere with the conduct of the study.
* Subject has current or past history of seizure disorder or brain injury, or any condition which, in the opinion of the investigator, predisposes to seizure; subject treated with other medications or treatment regimens that lower seizure threshold; subject undergoing abrupt discontinuation of alcohol or sedatives (including benzodiazepines)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08-06 (Actual); Primary Completion 2007-10-11 (Actual); Study Completion 2007-10-11 (Actual)

PRIMARY OUTCOMES:
Bioavailability and maximal concentration of the drug measured between 0 hours and 216 hours post dose. | measured between 0 hours and 216 hours post dose

SECONDARY OUTCOMES:
Time to maximal concentration measured between 0-216h post dose. Clinically relevant changes from baseline in clinical laboratory parameters (48 hours post dose), ECGs (0-48h post dose) and vital signs (0-48 hours post dose and any AEs during the study. | Time to maximal concentration measured between 0-216h post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Results for study 109169 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NAP109169?search=study&search_terms=109169#rs